CLINICAL TRIAL: NCT00085436
Title: A Phase II Study Of Autologous Tumor/DC Vaccine (DC Vaccine) Combined With Interleukin-2 (IL-2) And Interferon-α-2a (IFNα-2a) In Patients With Metastatic Renal Cell Carcinoma (RCC)
Brief Title: DC Vaccine Combined With IL-2 and IFNα-2a in Treating Patients With mRCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0238; R01CA095648 (NIH); P30CA023108 (NIH); DMS-0238 (Other: Dartmouth College); DMS-16090 (Other: Dartmouth College)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2013-06-10 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-05

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — aldesleukin; Interleukin-2; chiron; FANG vaccine; lentiviral minigene vaccine of COVID-19 coronavirus; Interferon-alpha; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccine, Aldesleukin-2, Interferon-a (Experimental): All patients will be treated with autologous tumor cell vaccine administered into inguinal lymph nodes via ultrasound guidance in addition to systemic IL-2 and recombinant interferon alfa. Two cycles of induction IL-2/IFNα-2a followed by 3 cycles of maintenance IL-2 + IFNα-2a.
  Interventions: Biological: Aldesleukin,; Biological: autologous tumor cell vaccine; Biological: recombinant interferon alfa

INTERVENTIONS:
Biological: Aldesleukin, — Recombinant human interleukin-2 (Proleukin, Chiron Therapeutics) will be administered as a five day (120 hr) continuous intravenous infusion at a dose of 18x106 IU per square meter of body surface area per day as per the Negrier regimen (21). The treatment schedule consists of two induction cycles and three maintenance cycles. Each induction cycle consists of two five-day courses of interleukin-2 infusion separated by a nine-day break. Each maintenance cycle consists of a five-day infusion followed by 23-day rest period of no therapy.
  Other Names: IL-2 (Proleukin®, Chiron)
Biological: autologous tumor cell vaccine — we will administer 1 X 107 DC cells. The autologous tumor cell vaccine (1 X 107 cells/1cc) in lactated ringers solution and injected into one (or two if clinically necessary) inguinal lymph nodes under ultrasound guidance. Each cycle of DC vaccine will be administered alternately in the right and left inguinal lymph nodes.
  Other Names: DC Vaccine
Biological: recombinant interferon alfa — Recombinant human interferon alfa-2a (Roferon, Roche), at a dose of 6 million IU per day three times a week subcutaneously will be given during the two interleukin-2 induction cycles and during each interleukin-2 maintenance cycle
  Other Names: interferon alfa-2a; Roferon

SUMMARY:
RATIONALE: Vaccines made from a patient's dendritic cells and tumor cells may make the body build an immune response to kill tumor cells. Interleukin-2 may stimulate a person's lymphocytes to kill kidney cancer cells. Interferon alfa may interfere with the growth of cancer cells. Combining vaccine therapy with interleukin-2 and interferon alfa may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving vaccine therapy together with interleukin-2 and interferon alfa works in treating patients with metastatic renal cell carcinoma (kidney cancer).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the clinical response rate in patients with metastatic renal cell carcinoma treated with autologous dendritic cells (DC) loaded with autologous tumor lysate (DC vaccine) in combination with interleukin-2 and interferon-alfa.
* Determine the toxicity of this regimen in these patients.

Secondary

* Determine, within relevant immune pathways, the treatment-related, tumor-specific immune response in patients treated with this regimen.
* Correlate tumor-specific immune response with objective clinical response in patients treated with this regimen.

OUTLINE:

* Induction therapy: Patients undergo leukapheresis on day -9. Patients receive autologous dendritic cells (DC) loaded with autologous tumor lysate (DC vaccine) by intranodal injection on days 0 and 14; interleukin-2 (IL-2) IV continuously on days 1-5 and 15-19; and interferon-alfa (IFN-α) subcutaneously (SC) once daily on days 1, 3, 5, 15, 17, and 19.
* Maintenance therapy: Patients undergo leukapheresis on days 33, 61, and 89. Patients receive DC vaccine by intranodal injection on days 42, 70, and 98; IL-2 IV continuously on days 43-47, 71-75, and 99-103; and IFN-α SC once daily on days 43, 45, 47, 71, 73, 75, 99, 101, and 103.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 18-33 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic renal cell carcinoma with measurable disease.
* Tumor tissue available and properly stored for lysate preparation.
* Patients must be at least 4 weeks from their last immunotherapy, radiation, surgery or chemotherapy (6 weeks for nitrosureas) and recovered from all ill effects.
* Karnofsky Performance Status ≥60%
* Life expectancy ≥ twelve weeks
* Adequate end organ function:
* Hematological: ANC ≥ 1000cells/μL, platelets ≥ 75,000/μL, hemoglobin ≥ 8.5 g/dl
* Liver: AST < 2 x ULN (upper limit of normal) unless due to metastases then < 5 x ULN, serum total bilirubin < 2 x ULN (except for patients with Gilbert's Syndrome)
* Renal: serum creatinine < 2.0 x ULN.
* Pulmonary: FEV1 > 2.0 liters or > 75% of predicted for height and age.
* Cardiac: No evidence of congestive heart failure, symptoms of coronary artery disease, myocardial infarction less than 6 months prior to entry, or serious cardiac arrhythmias. Patients over 40 or have had previous myocardial infarction greater than 6 months prior to entry will be required to have a negative or low probability cardiac stress test for cardiac ischemia.
* CNS: No history of brain metastases.
* Women should not be lactating and, if of childbearing age, have a negative pregnancy test within two weeks of entry to the study.
* Appropriate Contraception in both sexes

EXCLUSION CRITERIA:

* Patients may have not have been treated previously with IL-2, IFNα or autologous vaccine.
* Concomitant second malignancy except for non-melanoma skin cancer, and non- invasive cancer such as cervical CIS, superficial bladder cancer without local recurrence, breast CIS.
* In patients with a prior history of invasive malignancy, less than five years in complete remission
* Positive serology for HIV, hepatitis B or hepatitis C,
* Significant co-morbid illness such as uncontrolled diabetes or active infection that would preclude treatment on this regimen.
* Use of corticosteroids or other immunosuppression (if patient had been taking steroids, at least 4 weeks must have passed since the last dose).
* History of autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2003-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc S. Ernstoff, MD, Study Chair — Norris Cotton Cancer Center
Locations (1):
- Norris Cotton Cancer Center at Dartmouth - Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Result] Schwaab T, Schwarzer A, Wolf B, Crocenzi TS, Seigne JD, Crosby NA, Cole BF, Fisher JL, Uhlenhake JC, Mellinger D, Foster C, Szczepiorkowski ZM, Webber SM, Schned AR, Harris RD, Barth RJ Jr, Heaney JA, Noelle RJ, Ernstoff MS. Clinical and immunologic effects of intranodal autologous tumor lysate-dendritic cell vaccine with Aldesleukin (Interleukin 2) and IFN-alpha2a therapy in metastatic renal cell carcinoma patients. Clin Cancer Res. 2009 Aug 1;15(15):4986-92. doi: 10.1158/1078-0432.CCR-08-3240. Epub 2009 Jul 21. PMID 19622576

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were 18 and older, had measurable disease and newly progressive metastatic or new metastatic disease, tumor tissue for vaccine preparation, and signed consent. Eighteen mRCC patients were enrolled between January 2004 and August 2006.
Groups:
- All Patients Treated With DC Vaccine: All patients treated with autologous peripheral blood mononuclear cell-derived dendritic cells (DC) loaded with autologous tumor lysate (termed DC vaccine) administered into inguinal lymph nodes via ultrasound guidance in addition to systemic IL-2 and IFNα-2a. Two cycles of induction IL-2/IFNα-2a followed by 3 cycles of maintenance IL-2 + IFNα-2a.
Period: Overall Study
Arm/Group | All Patients Treated With DC Vaccine
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment: All patients will be treated with autologous peripheral blood mononuclear cell-derived dendritic cells (DC) loaded with autologous tumor lysate (termed DC vaccine) administered into inguinal lymph nodes via ultrasound guidance in addition to systemic IL-2 and IFNα-2a. Two cycles of induction IL-2/IFNα-2a followed by 3 cycles of maintenance IL-2 + IFNα-2a.
Arm/Group | Treatment
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (9.83126)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response as Measured by RECIST
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: monthly, then every 2-3 months
Population: Clinical response as measured by RECIST monthly and then every 2-3 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Units Other Than Participants: Clinical Response
Arm/Group | Treatment
Number analyzed (Participants) | 18
Number analyzed (Clinical Response) | 18
percentage of participants | 50 [22 to 66]

2. Secondary Outcome: Immunity as Measured by T-cell and Antibody Responses to the Tumor
Description: All patients receiving at least one week of treatment and have at least two time points available for assessment of immune parameters will be include in the evaluation of immune status.
Time Frame: monthly for 5 months
Measure: Number (95% Confidence Interval); unit: pg/mL (picogram/milliliter)
Groups:
- Vaccine, Aldesleukin-2, Interferon-a: All patients will be treated with autologous tumor cell vaccine administered into inguinal lymph nodes via ultrasound guidance in addition to systemic IL-2 and recombinant interferon alfa. Two cycles of induction IL-2/IFNα-2a followed by 3 cycles of maintenance IL-2 + IFNα-2a.
  Characterization of lymphocyte sub population by flow cytometry.
Arm/Group | Vaccine, Aldesleukin-2, Interferon-a
Number analyzed (Participants) | 18
pg/mL (picogram/milliliter)
  IP-10 Pre treatment | 126 [55 to 197]
  IP-10 Post treatment | 521 [277 to 765]

ADVERSE EVENTS:
Time Frame: 2 years, 7 months
Description: no difference
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 18/18
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=18)
Pruritis (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 3
Hypotension (Cardiac disorders) | 5
Metabolic Changes (Metabolism and nutrition disorders) | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No